CLINICAL TRIAL: NCT00471003
Title: A Non-Interventional, Post-Marketing Surveillance Phase IV Study to Asses the Efficacy and Safety of Telmisartan, With the Special Attention on the Influence of Telmisartan on Selected Metabolic Parameters of Patients
Brief Title: The Real-Life Efficacy and Safety of Telmisartan in Patients With Arterial Hypertension
Acronym: METABOLIC
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Affairs Therapeutic Area Head, Bayer Sp. z o.o
Other Study IDs: 12729; KL0601PL; 13929 - KL0601SI; 12804 - KL0601SK; 14326 - KL0601HR; NCT00459095 (obsolete NCT alias)
Record Dates: First submitted 2007-05-07; First posted 2007-05-08 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Hypertension
Keywords: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Arm 1
  Interventions: Drug: Pritor (Telmisartan , BAY68-9291)

INTERVENTIONS:
Drug: Pritor (Telmisartan , BAY68-9291) — Primary care hypertensive patients starting the therapy with Telmisartan

SUMMARY:
The main purpose of this study is to asses the efficacy and safety of telmisartan, with the special attention on the influence of telmisartan on selected metabolic parameters of patients.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Untreated or ineffectively treated arterial hypertension

Exclusion Criteria:

* Cholestatic disorders and severe hepatic failure
* Allergy to telmisartan
* Pregnancy and lactation period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 5448 (Actual)
Dates: Start 2006-09; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Efficacy and safety of the treatment with telmisartan reported by the physician | At the both of planned control visits. (Approx. interval between visits 3 months)

SECONDARY OUTCOMES:
Changes in metabolic parameters in telmisartan treated patients | At the both of planned control visits. (Approx. interval between visits 3 months)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (4):
- Many Locations, Croatia
- Many Locations, Poland
- Many Locations, Slovakia
- Many Locations, Slovenia